CLINICAL TRIAL: NCT01285102
Title: Phase II Study of Drug-eluting Irinotecan Beads (DEBIRI) in Refractory Metastatic Colorectal Cancer With Liver-only or Liver-predominant Disease
Brief Title: Chemoembolization Using Irinotecan in Treating Patients With Liver Metastases From Metastatic Colon or Rectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed early by the DSMB due to increased toxicity.
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-002; NCI-2010-01114 (Other: Nation Cancer Institutes); GI-063 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Liver Metastases; Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The first cohort of patients will receive a dose of 50 mg of irinotecan per DEBIRI treatment. We will escalate by 25 mg with subsequent cohorts up to a dose of 100 mg of irinotecan per DEBIRI treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Arm I (Experimental): Patients receive irinotecan-eluting beads via hepatic artery embolization every 3 weeks for up to 3 (unilobar disease) or 4 (bi-lobar disease) courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Combination Product: irinotecan-eluting beads; Procedure: hepatic artery embolization

INTERVENTIONS:
Combination Product: irinotecan-eluting beads — Patients will be treated with drug-eluting irinotecan beads per protocol at up to 100 mg per dose every 3 weeks. Patients will receive chemoembolization using LC Bead, loaded with irinotecan. The beads size range used in the study will be 100-300µm (nominal) with a dose of up to 100mg irinotecan per treatment. The beads will be mixed with a non-ionic contrast media in the vial immediately prior to use according to the instructions for use. Irinotecan will be loaded onto the beads not more than 2 hours prior to the procedure. The study goal will be to deliver the full dose of 100mg of irinotecan per treatment
  Other Names: DEBIRI
Procedure: hepatic artery embolization — Using a unilateral femoral approach, selective catheterization of the hepatic artery will be performed. Vascular access is obtained via the common femoral artery and a guide-wire advanced under fluoroscopic guidance. A microcatheter is then inserted over the guide-wire. The superior mesenteric artery is selected and an angiogram performed to identify any aberrant arterial anatomy and verify antegrade portal vein flow. The celiac axis is then selected and an angiogram completed. The catheter and guide-wire are used to select the proper hepatic artery and a limited angiogram performed to identify the branches of the hepatic artery. The right or left hepatic artery is selected distal to the cystic artery (if visualized), depending on the location of the lesions to be treated. The LC Bead, loaded with irinotecan will be delivered into the artery.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Chemoembolization kills tumor cells by blocking blood flow to the tumor and keeping chemotherapy drugs near the tumor.

PURPOSE: This phase II trial is studying how well chemoembolization using irinotecan works in treating patients with liver metastases from metastatic colon or rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the response rate of colorectal liver metastases (in the treated lobe) treated with DEBIRI, in refractory mCRC patients.

SECONDARY OBJECTIVES:

I. To evaluate the time to progression in the treated lobe for this patient population.

II. To evaluate the overall survival for this patient population. III. To evaluate patient tolerance and the toxicity profile of treatment with DEBIRI in this patient population.

OUTLINE:

Patients receive irinotecan-eluting beads via hepatic artery embolization every 3 weeks for up to 3 (unilobar disease) or 4 (bi-lobar disease) courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic to the liver and for which standard curative measures do not exist
* Patients must have received prior irinotecan-based treatment for their disease and had documented progression by RECIST criteria; patients must also have received prior fluoropyrimidine and oxaliplatin-based therapy
* Liver disease must not be amenable to potentially curative surgical resection
* Patients must have liver-only or liver-predominant disease to be eligible for this study; hepatic disease must be dominant, but patients are allowed to have extrahepatic disease provided it is not judged likely to be life threatening within 3 months
* Patients must have a patent portal vein as documented by CT, MRI, or ultrasound
* Prior radiation therapy is allowed but must have been completed >= 4 weeks prior to study entry; patients with history of prior radiation to the liver including radio-labeled microspheres cannot take part in this study
* Eastern Cooperative Oncology Group performance status 0-1
* Previous surgery or RFA to the liver is allowed; patients with history of chemoembolization or radio-labeled microspheres are excluded
* Life expectancy of >= 12 weeks
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< ULN
* AST(SGOT)/ALT(SGPT)/Alkaline Phosphatase =< 2.5 X institutional ULN
* Creatinine < 2.0 mg/dL
* PT/PTT < 1.5 X ULN
* Women of childbearing potential (WOCBP) and sexually active males must agree to use an accepted and effective method of contraception prior to study entry and for the duration of the study; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal; even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy) should be considered to be of child bearing potential
* Patients must demonstrate ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy (including targeted therapy i.e. cetuximab, panitumumab) or radiotherapy =< 4 weeks or treatment with bevacizumab =< 6 weeks prior to entering the study or those who have not recovered from acute adverse events due to agents administered more than 4 weeks earlier, with the exclusion of alopecia or neuropathy; patient with history of radiation to the liver including radio-labeled microspheres at any point in their past will be excluded
* Patients may not be receiving nor have received any other investigational agent =< 4 weeks prior to study registration
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including death from the therapeutic agents
* Patients with known brain metastases are excluded from this study because of their poor prognosis and frequent development of progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events
* As patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, known HIV-positive patients and those with known hepatitis B or C are excluded from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active bacterial infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically evident ascites requiring medical management or paracentesis, or Childs-Pugh score B/C are not eligible
* Patients with evidence of other cancer within 5 years, excluding adequately treated basal cell carcinoma of the skin
* Patient with significant cardiac, renal or hematologic or pulmonary dysfunction
* Patients with previous chemoembolization to liver metastases
* Patients may not receive any other anticancer therapy while on study, including immunotherapy; patients may not receive any other clinical investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Dotan, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DEBIRI With Hepatic Artery Embolization: Patients receive irinotecan-eluting beads via hepatic artery embolization every 3 weeks for up to 3 (unilobar disease) or 4 (bi-lobar disease) courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | DEBIRI With Hepatic Artery Embolization
Started | 4
Completed | 0
Not Completed | 4
Not completed — Closed to accrual by sponsor due to poor accrual and challenge with dosing | 4

BASELINE CHARACTERISTICS:
Arm/Group | DEBIRI With Hepatic Artery Embolization
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 77.5 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Time Frame: Duration of time from start of treatment to progression
Population: Study was closed to accrual by sponsor due to poor accrual and challenge with dosing. No data was generated.
Arm/Group | DEBIRI With Hepatic Artery Embolization
Number analyzed (Participants) | 0

2. Primary Outcome: Patient Tolerance and Toxicity Profile
Time Frame: First treatment then 30 days after completion of treatment then every 3 months for 2 years
Population: Study was closed to accrual by sponsor due to poor accrual and challenge with dosing. No data was generated.
Arm/Group | DEBIRI With Hepatic Artery Embolization
Number analyzed (Participants) | 0

3. Primary Outcome: Overall Survival
Time Frame: 30 days after completion of treatment then every 3 months for 2 years
Population: Study was closed to accrual by sponsor due to poor accrual and challenge with dosing. No data was generated.
Arm/Group | DEBIRI With Hepatic Artery Embolization
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | DEBIRI With Hepatic Artery Embolization
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEBIRI With Hepatic Artery Embolization (N=4)
Elevated ALP (Gastrointestinal disorders) | 4
Elevated AST (Gastrointestinal disorders) | 4
Elevated ALT (Gastrointestinal disorders) | 4
Elevated bilirubin (Gastrointestinal disorders) | 3
Biliary obstruction (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT01285102/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT01285102/ICF_001.pdf